CLINICAL TRIAL: NCT03077906
Title: Study of Gastro-oesophageal Reflux in Patients Having Had Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Reflux
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroœsophageal Reflux; Sleeve Gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Existing gastroœsophageal reflux: Patients who benefited from a sleeve gastrectomy surgery between 2008 and the end of 2015 in the department of digestive surgery of the CHU Brugmann.
  Patients who already had a disabling gastroœsophageal reflux resistant to medical treatment in pre-op, and lost it in post-op.
  Interventions: Other: Medical Files data extraction
- De novo gastroœsophageal reflux: Patients who benefited from a sleeve gastrectomy surgery between 2008 and the end of 2015 in the department of digestive surgery of the CHU Brugmann.
  Patients who developped gastroœsophageal reflux de novo.
  Interventions: Other: Medical Files data extraction

INTERVENTIONS:
Other: Medical Files data extraction — Medical Files data extraction

SUMMARY:
Obesity surgery has become commonplace nowadays. This type of surgery is in full swing and although it is mostly beneficial for the health of the patient (reduction of cardiovascular risks, improvement of self image, reduction of osteo-articular risks, etc...) it is however associated with risks. There are several short and long term complications, excluding the ones related to the anesthesia and the post-op recovery: fistulas, abcesses, infections, dysphagia, risks of endobrachyoesophagus, etc...

The gastroœsophageal reflux remains by far the most common post-op complaint within patients. Patients can experience symptoms as far as 3 years after the surgery. Medical treatment alone can in most cases lighten the symptoms. However, in some cases, this treatment fails and another type of surgery (bypass) must be undertaken, which is psychologically traumatic for the patient.

This retrospective study will analyze a cohort of patients who underwent bariatric surgery (mainly sleeve gastrectomy), in order to identify those at risk of developping gastroœsophageal reflux and how this complication can be avoided in pre-op. The study will also identify cases of invalidating gastroœsophageal reflux that can be solved by obesity surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had at least 1 year of postoperative follow-up

Exclusion Criteria:

* Patients who did not have postoperative gastroœsophageal reflux
* Patients who stopped their postoperative follow-up
* Patients with unsufficient data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who benefited from a sleeve gastrectomy surgery between 2008 and the end of 2015 in the department of digestive surgery of the CHU Brugmann.
  Patients who already had a disabling gastroœsophageal reflux resistant to medical treatment in pre-op and lost it in post-op, or patients who developped a gastroœsophageal reflux de novo.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
date of birth | 8 years
  date of birth of the patient
pre-op BMI | 8 years
  BMI of the patient before the surgical intervention
post-op BMI | 8 years
  BMI of the patient after the surgical intervention
existing pre-op gastroœsophageal reflux | 8 years
  existing gastroœsophageal reflux before the surgical intervention
post-op gastroœsophageal reflux | 8 years
  gastroœsophageal reflux after the surgical intervention
occurence of other surgical interventions | 8 years
  occurence of other obesity surgical interventions
medical complications | 8 years
  occurence of medical complications
number of clips used during the surgery | 8 years
  number of clips used during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Wauthy, MD, Study Director — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nilsson M, Johnsen R, Ye W, Hveem K, Lagergren J. Obesity and estrogen as risk factors for gastroesophageal reflux symptoms. JAMA. 2003 Jul 2;290(1):66-72. doi: 10.1001/jama.290.1.66. PMID 12837713
- [Background] Mora F, Cassinello N, Mora M, Bosca M, Minguez M, Ortega J. Esophageal abnormalities in morbidly obese adult patients. Surg Obes Relat Dis. 2016 Mar-Apr;12(3):622-628. doi: 10.1016/j.soard.2015.08.002. Epub 2015 Aug 7. PMID 26686303
- [Background] Huseini M, Wood GC, Seiler J, Argyropoulos G, Irving BA, Gerhard GS, Benotti P, Still C, Rolston DD. Gastrointestinal symptoms in morbid obesity. Front Med (Lausanne). 2014 Dec 4;1:49. doi: 10.3389/fmed.2014.00049. eCollection 2014. PMID 25593922
- [Background] Pallati PK, Shaligram A, Shostrom VK, Oleynikov D, McBride CL, Goede MR. Improvement in gastroesophageal reflux disease symptoms after various bariatric procedures: review of the Bariatric Outcomes Longitudinal Database. Surg Obes Relat Dis. 2014 May-Jun;10(3):502-7. doi: 10.1016/j.soard.2013.07.018. Epub 2013 Aug 29. PMID 24238733
- [Background] DuPree CE, Blair K, Steele SR, Martin MJ. Laparoscopic sleeve gastrectomy in patients with preexisting gastroesophageal reflux disease : a national analysis. JAMA Surg. 2014 Apr;149(4):328-34. doi: 10.1001/jamasurg.2013.4323. PMID 24500799
- [Background] El-Hadi M, Birch DW, Gill RS, Karmali S. The effect of bariatric surgery on gastroesophageal reflux disease. Can J Surg. 2014 Apr;57(2):139-44. doi: 10.1503/cjs.030612. PMID 24666452